CLINICAL TRIAL: NCT02457013
Title: Interest of High Flow Nasal Cannula (HFNC) Versus Non Invasive Ventilation During the Initial Management of Severe Bronchiolitis in Infants
Acronym: TRAMONTANE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9433
Record Dates: First submitted 2015-01-27; First posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HFNC treatment (Experimental): HFNC : High flow nasal canula 24hours Patients will be treated by a High flow nasal canula (HFNC: 2l/kg/min) for the initial management of their bronchiolitis (24 hours)
  Interventions: Device: HFNC
- nCPAP treatment (Active Comparator): nCPAP : nasal NCPAP Patients will be treated by a nasal CPAP (n-CPAP: 7 cmH2O) for the initial management of their bronchiolitis (24 hours)
  Interventions: Device: nCPAP

INTERVENTIONS:
Device: HFNC — Hygh flow nasal canula HFNC
  Arms: HFNC treatment
Device: nCPAP — nasal nCPAP
  Arms: nCPAP treatment

SUMMARY:
1. The purpose of the study is to evaluate prospectively the clinical benefits of High flow nasal canula (HFNC: 2l/kg/min) versus nasal CPAP( continuous positive airway pressure) (n-CPAP: 7 cmH2O) in the initial management of bronchiolitis in infants.
2. Design: non-inferiority study, prospective, controlled, randomized, multi-center.
3. Design: Infants less than 6 month admitted in pediatric intensive care unit for respiratory distress (mWCAS >3) secondary to bronchiolitis but not requiring mechanical ventilation will be randomized in two groups: "n-CPAP"(nasal continuous positive airway pressure) or "HFNC" during 24 hours.
4. Conditions of measurements:

   Primary endpoint: Proportion of failure in both arms during the first 24 hours. Failure criteria: A raise of the Clinical score for respiratory distress (mWCAS) (1 point) or respiratory rate (10/min /H0 and above 60/min) or discomfort (EDIN) (1point /H0 and above 4) or apnea.

   Secondary outcomes: Assessment at H1, H12, H24 of mWCAS, respiratory and heart rate, EDIN score, skin lesions, FiO2 (fraction of inspired oxygen

   ) required to achieve an oxygen saturation between 94 and 97%, transcutaneous PCO2 (carbon dioxide partial pressure) (correlated to an initial gas analysis), Report SpO2 / FiO2
5. Statistic: Intention to treat Analysis. Expected number of patients: 71 per arm: 142 children.
6. Study Schedule: October 2014-April 2016

ELIGIBILITY:
Inclusion Criteria:

* age<6months
* bronchiolitis
* mWCAS > or=3
* hospitalisation in pediatric intensive care unit
* signed consent form (2 parents)

Exclusion Criteria:

* Intubated patient
* Neurological or cardiac disease

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of failure | 24 hours
  Proportion of failure in both arms during the first 24 hours. A raise of the Clinical score for respiratory distress (mWCAS) (1 point) or respiratory rate (10/min /H0 and above 60/min) or discomfort (EDIN) (1point /H0 and above 4) or apnea.

SECONDARY OUTCOMES:
number of participants with an aggravation of the clinical score for respiratory distress arms | 1hour
  comparison of the clinical score for respiratory distress (mWCAS) in both arms
number of participants with an aggravation of the clinical score for respiratory distress arms | 12hours
  comparison of the clinical score for respiratory distress (mWCAS) in both arms
number of participants with an increase of the clinical score for respiratory distress arms | 1 hour
  Assessment of Report Sp02/Fi02in both arms
Comparison of the Report Sp02/Fi02 in both arms | 1 hour
  Assessment of Report Sp02/Fi02in both arms
Comparison of the Report Sp02/Fi02 in both arms | 12 hours
  Assessment of Report Sp02/Fi02in both arms
Comparison of the Report Sp02/Fi02 in both arms | 24 hours
  Assessment of Report Sp02/Fi02in both arms
number of participants with skin lesions in both arms | 1 hour
  number of participants with skin lesions in both arms and classification of the lesions with the National Pressure Ulcer Advisory Panel (NPUAP)
number of participants with skin lesions in both arms | 12 hours
  number of participants with skin lesions in both arms and classification of the lesions with the National Pressure Ulcer Advisory Panel (NPUAP)
number of participants with skin lesions in both arms | 24 hours
  number of participants with skin lesions in both arms and classification of the lesions with the National Pressure Ulcer Advisory Panel (NPUAP)
number of participants with Discomfort in both arms | 1 hour
  Assessment of the discomfort in both arms with the score of EDIN
number of participants with Discomfort in both arms | 12 hours
  Assessment of the discomfort in both arms with the score of EDIN
number of participants with Discomfort in both arms | 24 hours
  Assessment of the discomfort in both arms with the score of EDIN

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France